CLINICAL TRIAL: NCT04173364
Title: Interscalene Block and Dysfunction Diaphragmatic: Effect of Low Volume of Ropivacaine 0,1%. A Randomised, Controlled Trial
Brief Title: Interscalene Block and Dysfunction Diaphragmatic
Acronym: NUMEROBIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018_66; 2019-001984-62 (EudraCT Number)
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Diaphragmatic Paralysis
Keywords: interscalene block; shoulder surgery; local anesthesic; respiratory function; diaphragmatic dysfunction; echography; locoregional anesthesia
MeSH Terms: conditions — Respiratory Paralysis; Respiratory Aspiration | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : ropivacaine 0.1% (Experimental): Interscalene block for arthroscopic shoulder surgery with small volume of low concentration (0.1%) of ropivacaine
  Interventions: Drug: Ropivacaine 0.1% Injectable Solution
- control group : ropivacaine 0.5% (Active Comparator): Interscalene block for arthroscopic shoulder surgery with small volume of standard concentration (0.5%) of ropivacaine
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.5% Injectable Solution — Injectable solution of ropivacaine 0.5%
  Other Names: naropeine 0.5%
  Arms: control group : ropivacaine 0.5%
Drug: Ropivacaine 0.1% Injectable Solution — Dilution of ropivacaine to the concentration of 0.1%
  Other Names: Naropeine 0.1%
  Arms: Experimental group : ropivacaine 0.1%

SUMMARY:
The study seeks to show that interscalene injection of a small volume (<8ml) of ropivacaine at a low concentration (0.1%) reduces the frequency of hemi-diaphragmatic paresis compared to low volume injection at the standard concentration (0.5%) in patients undergoing arthroscopic shoulder surgery with ISB.

DETAILED DESCRIPTION:
It's a prospective monocentric randomized controlled clinical trial in 2 parallel groups in double blind.

the study concerns patients undergoing arthroscopic shoulder surgery with ISB. The study seeks to show that interscalene injection of a small volume (<8ml) of ropivacaine at a low concentration (0.1%) reduces the frequency of hemi-diaphragmatic paresis compared to low volume injection at the standard concentration (0.5%) in patients undergoing arthroscopic shoulder surgery with ISB.

Randomization in one of the two arms:

* Experimental group: <8ml ropivacaine 0.1%.
* Control group: <8mL of ropivacaine 0.5%.

Evaluation of diaphragmatic stroke by ultrasound and ventilatory function by spirometry and snip test before performing the ISB, then after installation of the ISB.

Performing the surgical procedure under general anesthesia assessment of postoperative analgesia and patient satisfaction during the following 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* orthopedic surgery compatible with interscalene block
* french speaking
* Patient who signed consent to participate in the study

Exclusion Criteria:

* Pregnant woman
* ASA score > 3
* Severe chronic respiratory insufficiency
* COPD >3 or 4 of Gold score
* coagulation trouble
* Allergic to medication involved in the study
* Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Compare the occurrence of hemi-diaphragmatic paresis | 1h after interscalene block
  Hemi diaphragmatic paresis is evaluated by quantifying the homolateral diaphragmatic stroke at interscalene block (ISB) by ultrasound analysis (measured in centimeter), during slow and deep inspiration. Diaphragmatic hemiparesis is defined as a decrease (at post-ISB time vs. pre-ISB time) of more than 25% of the diaphragmatic stroke during this slow and deep inspiration.

SECONDARY OUTCOMES:
Compare the frequency of hemi-diaphragmatic paralysis | 1h after interscalene block
  Hemi-diaphragmatic paralysis refers to the absence of diaphragmatic movement (or paradoxical movement) in ultrasound during rest ventilation and slow, deep inhalation.
Compare intraoperative analgesia | peroperative time
  Total consumption of sufentanil, and Analgesia Nociception Index values (ANI, MetroDoloris, France).
Compare postoperative analgesia | 24 hours postoperatively
  Duration of effective analgesia (defined as the period up to the first EVA > 3 (excluding PACU Consumption of morphine in PACU and analgesics within the first 24 hours.
Compare the ventilatory function (spirometry and snip test). | 1h after interscalene block
  Presence of a respiratory impairment detected by spirometry (Spiro-USB® device) and presence of a diaphragmatic impairment detected by snip test, (micro-RPM®). Ventilation impairment will be considered present if there is a decrease of at least 25% in vital capacity between the pre and post ISB. Diaphragmatic damage is defined as a decrease of at least 25% in the Snip-test values between the pre and post ISB.
Compare patient satisfaction | 24 to 48 hours postoperatively
  Evaluation of patient satisfaction by questionnaire at the patient's bedside or by telephone call within 24h-48h postoperatively. It is assessed on a numerical scale from 0 to 10 (0 being the lowest satisfaction value and 10 the highest value)
Compare the contralateral diaphragmatic stroke | 1h after interscalene block
  Evaluation of contralateral diaphragmatic compensation (diaphragmatic stroke in ultrasound, comparison of post-ISB time vs. pre-ISB time, expressed in %).

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud ALLUIN, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France